CLINICAL TRIAL: NCT01458834
Title: Attentional Training for Smoking Cessation Via Handheld Device or Personal Computer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Samantha Moshier, M.A., Principal Investigator, Boston University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BU-2453
Record Dates: First submitted 2011-10-22; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Smoking
Keywords: Smoking; Attentional bias; Craving
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active attention training condition (Experimental)
  Interventions: Behavioral: Attention bias modification task
- Control condition (Placebo Comparator)
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Attention bias modification task — Participants will complete a computerized probe-discrimination task from their home computer or handheld electronic device 3 times per day for one week. Each training session will consist of 160 trials. In each trial, two pictures (smoking-related or neutral) will appear on the screen simultaneously and then disappear. An arrow will appear in the location of one of the pictures (< or >). Participants are asked to quickly identify the direction of the arrow by pressing a button. In the active training task, the arrow will replace the neutral pictures 80% of the time.
  Arms: Active attention training condition
Behavioral: Control Condition — Participants will complete a computerized probe-discrimination task from their home computer or handheld electronic device 3 times per day for one week. Each training session will consist of 160 trials. In each trial, two pictures (smoking-related or neutral) will appear on the screen simultaneously and then disappear. An arrow will appear in the location of one of the pictures (< or >). Participants are asked to quickly identify the direction of the arrow by pressing a button. In the control training task, the arrow will replace the neutral and smoking-related pictures with equal frequency.
  Arms: Control condition

SUMMARY:
Several studies indicate that cigarette smokers show an attentional bias for cigarette-related cues, meaning that they more quickly detect and attend to and have more difficulty disengaging in cigarette-related information than neutral information. This bias is associated with craving and relapse following attempts to quit. This experiment will examine whether a computerized attentional training procedure will successfully reduce attentional bias towards smoking cues and reduce craving in regular cigarette smokers. The attentional training will be administered in a novel format in which participants complete 5-minute long training sessions 3 times per day and can complete the trainings via home computer or handheld device such as the iPhone, Android phone, or iPod touch. A baseline assessment in the laboratory will measure attentional bias to smoking cues and craving following smoking cue exposure. Participants will then be randomly assigned to either the active training condition or a control condition. In both conditions, participants will be asked to complete brief training sessions 3 times daily for one week using their personal computer or handheld device. Following one week of training, participants will return to the lab for endpoint assessment of attentional bias and craving. The investigators hypothesize that compared to the control condition, the active training condition will significantly reduce attentional bias toward smoking related cues and cue-induced cigarette craving.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65.
2. Familiarity with a computer keyboard and mouse.
3. Must own a iPhone, iPod Touch, or Google Android-based phone (such as the Droid or Nexus One) or have regular access to the Internet via personal computer.
4. Current regular smoker, as defined by self-reported use of at least 1 year and a current average of at least 10 cigarettes smoked per day.

Exclusion Criteria:

1. Individuals with current suicidality (determined by a score of 2 or 3 on item 9 of the Beck Depression Inventory given following consent) will be excluded from further participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Brief Questionnaire of Smoking Urges (QSU-Brief) | Assessed at baseline and endpoint visits (one week apart)
Attentional Bias Scores | Assessed at baseline and endpoint visits (one week apart)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Moshier, MA, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States